CLINICAL TRIAL: NCT02192645
Title: The Efficacy and Safety of Sanfujiu on Patients With Persistent Allergic Rhinitis: Randomized Controlled Study (SPAR Study)
Brief Title: The Efficacy and Safety of Sanfujiu on Patients With Persistent Allergic Rhinitis: Randomized Controlled Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Doctor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPAR
Record Dates: First submitted 2014-07-07; First posted 2014-07-17 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sanfujiu (Experimental): Formula for Sanfujiu: Huangjiezi; Xixin; Yanhusuo; and so on Acupoint for Sanfujiu: Different ten acupoints determined according to Chinese medicine theory for each time.
  Timepoint: Five times of 3 years at Sanfu Point application: The patients will be treated with herbal cake-separated moxibustion on acupoints and lasted 60 minutes each time.
  Interventions: Drug: Sanfujiu
- placebo (Placebo Comparator): Formula for placebo: Fuxiaomai; and so on. the appearance is similar as drugs of Sanfujiu Acupoint for placebo: Ten acupoints determined according to Chinese medicine theory are the same as Sanfujiu group of each timepoint .
  Timepoint: Five times per year for 3 years. Point application: The patients will be treated with placebo on acupoints and lasted 60 minutes each time.
  Interventions: Drug: Placebo
- waiting list (No Intervention): No intervention in the first year. Accept Sanfujiu in the second and the third years.

INTERVENTIONS:
Drug: Sanfujiu
  Other Names: Sanfu-moxibustion
  Arms: Sanfujiu
Drug: Placebo — The placebo ointment is composed of flour, buckwheat flour, food colorants and water, resulting in an ointment similar in appearance to the Sanfujiu ointment.
  Other Names: Placebo ointment
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether Sanfujiu is effective and safe in the treatment of persistent allergic rhinitis.

DETAILED DESCRIPTION:
The trial consists of 5 treatment sessions along with a one-year follow-up. This process is then repeated in the second and third years. Eligible participants diagnosed with PAR were randomized at a ratio of 2:2:1 into one of three groups: (a) SHP group; (b) placebo group; or (c) waiting-list group. The waiting-list group will receive no treatment in the first year, but will receive SHP in the following two years. The primary outcome, total nasal symptoms score, is self-assessed at the beginning of each treatment session and during each annual follow-up. Secondary outcomes include the Rhinoconjunctivitis Quality of Life Questionnaire, allergic rhinitis attacks, and relief medications. The trial will be stopped if early termination criteria are met during the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 with PAR, defined clinically as symptoms being present at least 4 days a week, for at least 4 weeks
* Test positive for allergen specific immunoglobulin E . Allergens include: mites (Dermatophagoides pteronyssinus and Dermatophagoides farinae), cockroach (Blatella germanica) and/or house dust
* Informed consent
* TNSS ≥3

Exclusion Criteria:

* Seasonal or chronic instance of other forms of rhinitis (i.e. sinusitis)
* Asthma and/or moderate to severe atopic dermatitis
* Allergy treatment at present due to asthma, eczema, atopic dermatitis, or other diseases
* Nasal structural abnormalities
* Severe mental illness, severe chronic respiratory diseases, severe diseases of the cardiovascular system, severe kidney disease, severe liver disease, severe blood system diseases, severe neurological and neuromuscular disease, severe metabolic and endocrine system disease, severe diabetes, immune function (including the application of immunosuppressant or HIV infection to low immune function etc.); The laboratory test indexes more than twice the upper limit of normal reference value or abnormal results that don't fit for the study confirmed by researchers;
* Blood coagulation dysfunction or patients are using anticoagulants
* Systemic corticosteroids treatment six months before the start of the study, or intranasal corticosteroids 15 days before the start of the study;
* Immunotherapy for more than 3 years;
* Alternative therapies such as acupuncture, traditional Chinese medicine (TCM) one month before the start of the study,or prepare to use during the study;
* Moxibustion therapy half years before the start of the study;
* Patients participating other clinical trials;
* Prepare to pregnancy, pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total nasal symptom score at 12 months | 12 months after treatment

SECONDARY OUTCOMES:
Change from baseline in Rhinitis Quality of Life Questionnaire at 12 months | 12 months after treatment
Responder rate of Rhinitis Quality of Life Questionnaire | 12 months after treatment
  Responders to study intervention are defined as patients with a change in Rhinitis Quality of Life Questionnaire score of ≥0.5 between the baseline and 12 months
The number of days of allergic rhinitis attack | 12 months after treatment
The quantity of conventional relief medication used | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjian Lu, Doctor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen X, Lu C, Stalsby-Lundborg C, Li Y, Li X, Sun J, Ouyang W, Li G, Su G, Lu L, Fu W, Wen Z. Efficacy and Safety of Sanfu Herbal Patch at Acupoints for Persistent Allergic Rhinitis: Study Protocol for a Randomized Controlled Trial. Evid Based Complement Alternat Med. 2015;2015:214846. doi: 10.1155/2015/214846. Epub 2015 Aug 2. PMID 26300945